CLINICAL TRIAL: NCT00225524
Title: Phase III Long-Term Administration Study of Effexor XR for the Treatment of Depression
Brief Title: Study Evaluating Long-Term Safety of Effexor XR in Patients With Major Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0600B1-818
Record Dates: First submitted 2005-09-12; First posted 2005-09-23 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Effexor XR

SUMMARY:
Phase III long-term safety study of Effexor XR in patients with major depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complete the Phase III double-blind study (Protocol Number 0600B1-816)

Exclusion Criteria:

* Patients with schizophrenia or any other psychotic disorder
* Patients with history or presence of bipolar disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-09

PRIMARY OUTCOMES:
Incidence of adverse events

SECONDARY OUTCOMES:
Quantitative data for laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (44):
- Japan (44):
  - Nagoya, Aichi-ken
  - Ichikawa, Chiba
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Ohnojyo, Fukuoka
  - Hiroshima, Hiroshima
  - Kure, Hiroshima
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Tsuchiura, Ibaragi
  - Tsukuba, Ibaragi
  - Kanazawa, Ishikawa-ken
  - Hanamaki, Iwate
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Kikuchi, Kumamoto
  - Nagasaki, Nagasaki
  - Ohmura, Nagasaki
  - Kashihara, Nara
  - Jyo-etsu, Niigata
  - Beppu, Ohita
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Sayama, Osaka
  - Saitama, Saitama
  - Hamamatsu, Shizuoka
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Kodaira, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Nakano-ku, Tokyo
  - Ohta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku, Tokyo
  - Tachikawa, Tokyo
  - Toshima-ku, Tokyo